CLINICAL TRIAL: NCT05976165
Title: Breath Testing for Small Intestinal Bacterial Overgrowth in Patients Treated With Proton Pump Inhibitors
Brief Title: A Study of Breath Testing for Small Intestinal Bacterial Overgrowth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andree H. Koop, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-007268
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastroesophageal Reflux; Regurgitation; Heartburn
Keywords: Proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breath Test Evaluation for SIBO (Experimental): Subjects with symptoms of gastroesophageal reflux disease (GERD) treated with a short course of proton pump inhibitors (PPI) clinically will undergo breath testing evaluating for small intestinal bacterial overgrowth (SIBO).
  Interventions: Other: Breath Testing

INTERVENTIONS:
Other: Breath Testing — Subjects drink a small carbohydrate solution, and then provide a breath sample every 15 minutes for one hour, and then every 30 minutes for the next two hours

SUMMARY:
Researchers hope to determine how often small intestinal bacterial overgrowth occurs after taking proton pump inhibitors.

ELIGIBILITY:
Inclusion criteria:

* Predominant symptoms of gastroesophageal reflux disease including heartburn, regurgitation
* Subjects must be able to give appropriate informed consent

Exclusion criteria:

* Prior diagnosis of SIBO
* Use of PPIs or H2R-anatagonstists in the prior 3 months
* Major concomitant illness (renal, hepatic, rheumatologic or cardiovascular disease, or malignancy)
* Antibiotic therapy within one month
* Prior gastrointestinal surgery including esophageal, gastric, and small or large bowel surgery
* Previously diagnosed irritable bowel syndrome or inflammatory bowel disease
* Individuals who are pregnant or breast feeding
* Patients with plans to become pregnant
* Inability to take PPIs, including allergy/sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of SIBO after treatment with PPI | After PPI therapy, approximately 8 weeks
  Number of subjects to have a positive breath testing for small intestinal bacterial overgrowth (SIBO) after clinical treatment of proton pump inhibitors (PPI ).

SECONDARY OUTCOMES:
Symptoms of SIBO after treatment with PPI | After PPI therapy, approximately 8 weeks
  Measured using the self-reported Mayo Bloating Questionnaire to assess symptoms of bloating and abdominal distension. Comprised of 45 questions addressing symptoms of bloating/distention. Other questionnaires include a diarrhea survey and the GERDQ.
Incidence of SIBO before treatment with a PPI | Baseline
  Number of subjects to have a positive breath testing for small intestinal bacterial overgrowth (SIBO) before clinical treatment of proton pump inhibitors (PPI ).
Symptoms of SIBO before treatment with a PPI | Baseline
  Measured using the self-reported Mayo Bloating Questionnaire to assess symptoms of bloating and abdominal distension. Comprised of 45 questions addressing symptoms of bloating/distention. Other questionnaires include a diarrhea survey and the GERDQ.

CONTACTS AND LOCATIONS:
Overall Officials: Andree Koop, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No